CLINICAL TRIAL: NCT01856166
Title: Programmed Intermittent Epidural Bolus Coupled With PCEA (PIEB-PCEA) Versus Continuous Epidural Infusion Coupled With PCEA (CEI-PCEA) for Labor Analgesia in Nulliparous: Effects on Labor Outcomes
Brief Title: PIEB-PCEA Versus CEI-PCEA for Labor Analgesia in Nulliparous
Acronym: PIEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 9147
Record Dates: First submitted 2013-04-29; First posted 2013-05-17 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy
Keywords: Nulliparous; Singleton; delivery; pregnancy
MeSH Terms: interventions — Levobupivacaine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CEI-PCEA (Active Comparator): Continuous Epidural Infusion coupled with Patient Controlled Epidural Analgesia
  Interventions: Device: Release analgesia by CADD SMITHS PCEA pump; Drug: Levobupivacaine; Drug: Sufentanil
- PIEB-PCEA (Experimental): Programmed Intermittent Epidural Bolus coupled with Patient Controlled Epidural Analgesia
  Interventions: Device: Release analgesia by CADD SMITHS PIEB pump; Drug: Levobupivacaine; Drug: Sufentanil

INTERVENTIONS:
Device: Release analgesia by CADD SMITHS PCEA pump — Analgesia will be release by continuous manner with an automatic pump
  Arms: CEI-PCEA
Device: Release analgesia by CADD SMITHS PIEB pump — Analgesia will be release by bolus with an automatic pump
  Arms: PIEB-PCEA
Drug: Levobupivacaine
Drug: Sufentanil

SUMMARY:
Epidural analgesia still have an impact on obstetric outcomes and especially on instrumented delivery rates.

To assess the best maintainance regimen of epidural analgesia during labor the investigators plan to include 300 nulliparous in this multicenter randomized, double blind trial. The primary outcome will be a composite set of criteria that can lead to instrumented delivery. Secondary outcome will focus on analgesia motor block and satisfaction.

DETAILED DESCRIPTION:
Patients will be informed during the anaesthetic consultation and recruited at the beginning of the labor if they comply with inclusion criteria. Habitual proceedings of the placing and induction of epidural analgesia (Local Anaesthetics (AL): Levobupivacaine 0.100% 15mL Sufentanil 10µg). Patients who will not obtain at 30min a pain score < 1/10 will be excluded (epidural analgesia not functional). The upkeep of analgesia will be provided by an automatic pump and randomized in: classic pump and new pump. The mixture used will be the same in the 2 groups: Levobupivacaine 0.0100% + Sufentanil 0.5µg/mL. The classic pump administers AL with a continuous output (8mL/h)even though the new pump administers AL in bolus (8mL every hour; beginning 1h after the induction). The classic pump is a pump CADD SMITHS PCEA (Patient Controlled Epidural Analgesia) with the programming: continuous output 8mL/h; Additional bolus if necessary: 8mL; Maximal dose by hour: 24mL.

The new pump is a pump CADD SMITHS called PIEB (Programmed Intermittent Epidural Bolus) with the programming: intermittent bolus 8mL every hour; Additional bolus if necessary: 8mL; Ban period during 10min between patient bolus and automatic bolus; Maximal dose by hour: 24mL.

In case of the pain reappears and which is not calmed with 2 successive patient bolus, the anaesthetist will be called for the evaluation and administration of a doctor bolus if necessary (Levobupivacaine 0.125% 5mL associated with 50µg of Clonidine).

Collected data will be demographic data, data about the obstetrical labor proceedings, data about pain, motor block, maternal satisfaction, total quantity of administered analgesia, number of patient and doctor bolus wich are asked and administered and neonatal data.

Endpoints will be collected by a doctor in blind of the type of pump (the 2 pumps are the same extern aspect, only the intern programming is different).

In case of caesarean during the labor, patient will be excluded of the study. When a decision of extraction will be taken, patient will receive a bolus of AL according to the anaesthetist decision but not accounted for the dose calculation.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous patient with a spontaneous labor at full term, from a normal pregnancy, carrier a singleton in cephalic position, with a distension <4cm and eligible for an epidural analgesia
* Patient has signed informed consent
* Patient affiliated or beneficiary of a social medical insurance
* Patient aged between 18 and 44 years old

Exclusion Criteria:

* Morphinic administration before the care
* Anomaly of fetal cardiac rate
* Fetal or maternal anomalies wich don't allow to evaluate motor block
* Known uterine malformation
* Contraindications for thrusts for pregnancy
* Patient protected by law
* Patient under guardianship

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 304 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Occurence of a specific clinical criteria which can lead to a complication of the delivery | Up to 10 hours
  Specific clinical criteria are:
  * Type of posterior engagement
  * Type of posterior extrication
  * Duration of waiting at complete dilatation > 3 hours
  * Duration of expulsive efforts > 40 minutes
  * Foetal bradycardia < 100 BPM during 1 minute at least

SECONDARY OUTCOMES:
Instrumental delivery rate | up to 10 hours
Pain during the end of labor | up to 10 hours
Efficacity of epidural analgesia | up to 10 hours
Efficacity of epidural analgesia | up to 10 hours
  Efficacity of epidural analgesia is defined by a EVN score < 3 at several times of delivery.
Presence of motor block | Up to 10 hours
  Presence of motor block is estimated with Bromage and Straigh Raising leg scales.

CONTACTS AND LOCATIONS:
Overall Officials: Estelle MORAU, PhD, Principal Investigator — CHU Montpellier - Department of gynaecology and obstetric
Locations (4):
- France (4):
  - Hôpital Mère Enfant, Bron
  - CHU d'Estaing, Clermont-Ferrand
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - CHU of Montpellier, Montpellier

REFERENCES:
- [Derived] Morau E, Jaillet M, Storme B, Nogue E, Bonnin M, Chassard D, Benhamou D, Nagot N, Dadure C. Does programmed intermittent epidural bolus improve childbirth conditions of nulliparous women compared with patient-controlled epidural analgesia?: A multicentre, randomised, controlled, triple-blind study. Eur J Anaesthesiol. 2019 Oct;36(10):755-762. doi: 10.1097/EJA.0000000000001053. PMID 31335447